CLINICAL TRIAL: NCT06331702
Title: A Phase Ⅳ, Randomized, Controlled, Open-label, Immunogenicity Study of Vero Cell-derived Inactivated Japanese Encephalitis Vaccine (JEV-I) Co-administered With Measles-Mumps-Rubella Vaccine (MMR)
Brief Title: Immunogenicity of Japanese Encephalitis Vaccine Co-administered With Measles-Mumps-Rubella Vaccine (MMR)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Liaoning Chengda Biotechnology CO., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDBJEIV2023001
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Japanese Encephalitis; Measles; Mumps; Rubella
MeSH Terms: conditions — Encephalitis, Japanese; Measles; Mumps; Rubella | interventions — Measles-Mumps-Rubella Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (JEV-I and MMR co-administration group) (Experimental): Participants will receive 1 dose of JEV-I and 1 dose of MMR concurrently on Day 0, with each vaccine administered on a different side of the body, and a second dose of JEV-I 7-10 days later. Blood sampling will be performed on Day 0 and 30 days after the second dose of JEV-I.
  Interventions: Biological: Vero cell-drived inactive Japanese encephalitis vaccine; Biological: Measles-Mumps-Rubella Vaccine
- Group 2 (JEV-I administered separately) (Active Comparator): Participants will receive 2 doses of JEV-I (7-10 days apart). Blood sampling will be performed on Day 0 and 30 days after the second dose of JEV-I.
  Interventions: Biological: Vero cell-drived inactive Japanese encephalitis vaccine
- Group 3 (MMR administered separately) (Active Comparator): Participants will receive 1 doses of MMR. Blood sampling will be performed on Day 0 and Day 30.
  Interventions: Biological: Measles-Mumps-Rubella Vaccine

INTERVENTIONS:
Biological: Vero cell-drived inactive Japanese encephalitis vaccine — 0.5ml for each dose, manufactured by Liaoning Chengda Biotechnology CO., LTD, administered in the deltoid area of lateral arm by intramuscular injection.
  Other Names: JEV-I
  Arms: Group 1 (JEV-I and MMR co-administration group); Group 2 (JEV-I administered separately)
Biological: Measles-Mumps-Rubella Vaccine — 0.5ml for each dose (after dissolving), manufactured by Shanghai Institute of Biological Products CO., LTD, administered in the lower part of the deltoid area of lateral arm, by subcutaneous injection.
  Other Names: MMR
  Arms: Group 1 (JEV-I and MMR co-administration group); Group 3 (MMR administered separately)

SUMMARY:
This is a phase IV, randomized, controlled, open-label study proceed in healthy children aged 8 months in China. The primary objective is to demonstrate the immunogenicity of simultaneous administration of JEV-I and MMR is not inferior to that of separate administration, as measured by seroconversion rates and antibody titers against the four antigens. The secondary objective is to describe the safety of the vaccines when administered simultaneously or separately.

DETAILED DESCRIPTION:
According to current immunization programs in China, there is an overlap in the vaccination schedules for JEV-I and MMR. Children are recommended to receive 2 doses of JEV-I at 8 months of age, with an interval of 7-10 days. The MMR vaccine is also recommended for administration at 8 months of age. Administering JEV-I and MMR vaccines simultaneously at 8 months of age may facilitate adherence to vaccination programs, reduce the burden of medical treatment for parents and children who receive both vaccines separately, and improve the efficiency of vaccination work.

This is a phase IV, randomized, controlled, open-label study proceed in healthy children aged 8 months in China. The primary objective is to demonstrate the immunogenicity of simultaneous administration of JEV-I and MMR is not inferior to that of separate administration, as measured by seroconversion rates and antibody titers against the four antigens. The secondary objective is to describe the safety of the vaccines when administered simultaneously or separately.

The children aged 8 months who have not received any Japanese encephalitis vaccine or MMR (or vaccines containing related ingredients) will be recruited and randomly assigned to one of three study groups (1:1:1 ratio): Group 1, Group 2 and Group 3. Participants in Group 1 will receive JEV-I (dose 1) and MMR simultaneously for the first time. Participants in Group 2 will receive JEV-I only. Participants in Group 3 will receive MMR only.

Blood will be collected pre-vaccination (Day 0) and 30 days post vaccination to evaluate seroconversion rates and antibody titers against the four antigens.

After each vaccination, all participants will be observed at the clinical site for at least 30 minutes for immediate reactions and will be monitored for solicited adverse events (AEs) for 7 days post vaccination. All participants will be monitored for unsolicited AEs and serious adverse events within 30 days of post vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 8 months to <12 months at the time of enrollment
* Participants are able to provide valid identification documents of themselves and/or their legal guardian (entrusted person).
* Legal guardian of the participants can understand requirements and processes of the study, voluntarily agree to participate in the clinical trial, provide informed consent, accept all scheduled visits.

Exclusion Criteria:

* Axillary temperature >37.0 ℃ at the time of enrollment.
* Participating in another clinical trial or planning to participate in another clinical trial during the course of this trial.
* Previous receipt of the Japanese encephalitis vaccine or the measles-mumps-rubella vaccine (or a vaccine containing any of these components), or plan to receive other vaccines of the same type or composition during the trial period.
* History of measles, mumps, rubella, or Japanese encephalitis infection (confirmed by clinical, serological, or microbiological methods).
* Received blood or blood products within 3 months before enrollment.
* History of allergies to any component of the experimental vaccine, or severe allergies to other vaccine or drugs administered in the past, such as anaphylactic shock, laryngeal edema, henoch-schonlein purpura, thrombocytopenic purpura, arthur reaction, dyspnea, angioneuroedema, systemic rash and/or urticaria.
* History of attenuated live vaccine administration within 14 days prior to vaccination, or history of other non live vaccine administration within 7 days prior to vaccination.
* Acute febrile diseases (axillary body temperature ≥ 38.5 ℃) or in acute stage of chronic diseases, or taking antipyretics, analgesics, and anti-allergic agents within 3 days before vaccination.
* Primary or acquired immunodeficiency, such as human immunodeficiency virus infection (participants themselves or their mothers are infected with human immunodeficiency virus), systemic lupus erythematosus, guillain-barre syndrome, or other autoimmune diseases.
* Primary or acquired immune dysfunction (history of thyroid, pancreatic, liver, and spleen resection)
* Receipt of immunosuppressive therapy within 3 months prior to enrollment, such as cytotoxic therapy, steroid therapy (defined as continuous oral or intravenous infusion for more than 14 days, with a glucocorticoid dose of ≥0.5 mg/kg/day, unrestricted for inhaled and local steroids), or long-term other immunomodulatory drugs.
* Serious illness (acute or chronic), known or suspected, such as complicated diabetes, infectious, purulent, and allergic skin diseases, Down's syndrome, sickle cell anemia, cardiovascular and cerebrovascular diseases, liver and kidney diseases, respiratory diseases, malignant tumors, etc.
* Contraindications to intramuscular injection, such as diagnosed with thrombocytopenia, any coagulation disorders, or receiving anticoagulant treatment.
* History of convulsions, epilepsy, encephalopathy, mental illness or other neurological disorders, or a family history of mental illness.
* Plans to move out of the local area before the end of the experiment or leave the local area for a long time during the scheduled trial visit period.
* Any conditions that may interfere with the evaluation of the experimental purpose, as deemed by the researcher.

Ages: 8 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 408 (Actual)
Dates: Start 2024-03-02 (Actual); Primary Completion 2025-02-11 (Actual); Study Completion 2025-02-11 (Actual)

PRIMARY OUTCOMES:
Antibody Titer for Post Vaccination | 30 days after the last dose of vaccination
  The serum neutralizing antibody titer against Japanese encephalitis virus is measured by plaque reduction neutralization test (PRNT). The immunoglobulin (IgG) antibody titers against measles virus, mumps virus, and rubella virus are measured using enzyme-linked immunosorbent assay (ELISA).
Seroconversion Rate for Post Vaccination | 30 days after the last dose of vaccination
  The seroconversion rate for JEV-I post vaccination is defined as the percentage of participants with a change in serum anti-JE neutralizing antibody from PRNT titer <1:10 at baseline to titer ≥1:10 30 days after the last dose of vaccination or a 4-fold rise from baseline. The seroconversion rate for MMR post vaccination is defined as the percentage of participants with a change in serum measles IgG antibody from titer <200 milli international units (mIU)/mL at baseline to titer ≥200 mIU/mL post vaccination or a 4-fold rise from baseline, and serum mumps IgG antibody from titer <100 international units (IU)/mL to titer ≥100 IU/mL or a 4-fold rise from baseline, and serum rubella IgG antibody from titer <20 IU/mL to titer ≥20 IU/mL or a 4-fold rise from baseline, as measured by ELISA.

SECONDARY OUTCOMES:
Incidence of Any Local and Systemic Adverse Events Within 30 Minutes of Each Vaccination | 30 minutes following each vaccination
  Participants will be observed at the clinical site for 30 minutes after each dose of vaccine. Any adverse events at the vaccination site (local) and non vaccination site (systemic) are collected. Adverse Events (AEs) are defined as all adverse medical events that occur in participants after receiving the investigational drug, which can manifest as symptoms, signs, diseases, or abnormal laboratory tests, but may not necessarily have a causal relationship with the investigational drug.
Incidence of Solicited Local and Systemic Adverse Events Within 7 Days of Each Vaccination | 30 minutes through 7 days following each vaccination
  Parents use a structured diary card to record the following solicited (pre-listed) local and system reactions from 30 minutes through 7 days following vaccination:
  Local reactions:
  * Induration
  * Swelling
  * Rash
  * Tenderness
  Systemic reactions:
  * Fever
  * Diarrhea
  * Constipation
  * Dysphagia
  * Anorexia
  * Sickness
  * Vomiting
  * Syncope
  * Convulsions
  * Cough
  * Pruritus
  * Irritability or Sleepiness
  * Skin and mucosal abnormalities
  * Fatigue
  * Acute Allergic Reactions
Incidence of Unsolicited Adverse Events and Serious Adverse Events Within 30 Days of Post Vaccination | 30 days of post vaccination
  Unsolicited adverse events and serious adverse events within 30 days of post vaccination will be collected through a combination of telephone visits by researchers and active reporting by participants.
  Serious adverse events are those meeting one of the following conditions:
  * Death
  * Life threatening
  * Resulted in a persistent or significant disability or incapacity
  * Required inpatient hospitalization or prolongation of existing hospitalization.
  * Congenital abnormalities or birth defects.

CONTACTS AND LOCATIONS:
Overall Officials: Huanyu Wang, Study Director — Liaoning Chengda Biotechnology CO., LTD
Locations (1):
- Jiangsu Provincial Center for Disease Control and Prevention, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No